CLINICAL TRIAL: NCT06413680
Title: A Phase 1/2a, Open-Label, Dose Escalation and Dose Expansion First-In-Human Study of the Safety, Tolerability, Activity, and Pharmacokinetics of REGN10597 (Anti-PD-1-IL-2RA-IL-2 Fusion Protein) Alone or in Combination With Cemiplimab in Patients With Advanced Solid Organ Malignancies
Brief Title: A First-In Human (FIH) Study to Find Out How Well REGN10597 Medicine Given Alone or in Combination With Cemiplimab Works in Adult Participants Who Have Cancer With Tumors That Have Spread in Their Body
Acronym: BrILliance
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R10597-ONC-22114; 2025-523399-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Melanoma; Clear-Cell Renal-Cell Carcinoma (ccRCC); Advanced Solid Tumors
Keywords: Advanced solid organ malignancies; Locally advanced; Metastatic; Non-uveal; Unresectable; Primary or secondary resistance to programmed cell death protein 1 (PD-1)/ programmed cell death ligand 1 (PD-L1)
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Monotherapy Dose Escalation (Experimental): Multiple Dose Level (DL) Cohorts to identify the Recommended Phase 2 Dose (RP2D)
  Interventions: Drug: REGN10597
- Phase 2: Monotherapy Dose Expansion (Experimental): Cohort 1: Melanoma participants Cohort 2: Clear-cell Renal-Cell Carcinoma (ccRCC) participants
  Interventions: Drug: REGN10597
- Phase 1: Combination Dose Escalation (Experimental): Multiple DL Cohorts to identify the RP2D
  Interventions: Drug: REGN10597; Drug: Cemiplimab
- Phase 2: Combination Dose Expansion (Experimental): Cohort 1: Melanoma participants
  Interventions: Drug: REGN10597; Drug: Cemiplimab

INTERVENTIONS:
Drug: REGN10597 — Administered per the protocol
Drug: Cemiplimab — Administered per the protocol
  Arms: Phase 1: Combination Dose Escalation; Phase 2: Combination Dose Expansion

SUMMARY:
This study is researching an experimental drug called REGN10597 alone or in combination with another drug called cemiplimab (called "study drug(s)"). The study is focused on patients with certain solid tumors that are in an advanced stage.

The aim of the study is to see how safe, tolerable, and effective the study drug(s) are.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug(s)
* How much study drug(s) is in the blood at different times
* Whether the body makes antibodies against the study drug(s) (which could make the study drug(s) less effective or could lead to side effects)

DETAILED DESCRIPTION:
Phase 1: Conducted in the United States only Phase 2: Conducted globally

ELIGIBILITY:
Key Inclusion Criteria:

Dose escalation cohorts:

1. Histologically or cytologically confirmed diagnosis of solid malignancy (locally advanced or metastatic) with confirmed progression on standard-of-care therapy
2. Participants are required to submit archival tissue if it is available

Dose expansion cohorts:

1. Histologically of cytologically confirmed diagnosis of one of the following tumors with criteria, as defined in the protocol:

   * Module 1, Cohort 1: anti-PD-(L)1 Progressed Melanoma or
   * Module 1, Cohort 2: anti-PD-(L)1 Progressed RCC or
   * Module 2, Cohort 1: 1L Melanoma
2. ALL Participants ARE REQUIRED to submit fresh pretreatment biopsy during screening, with an additional exploratory biopsy at other time points

Key Exclusion Criteria:

1. Prior treatment with Interleukin 2 (IL2)/IL15/IL-7 given outside the context of concurrent administration with adoptive cell therapy
2. Prior treatment with anti-PD1/PD-L1, or an approved systemic therapy or any previous systemic non-immunomodulatory biologic therapy within 4 weeks, as defined in the protocol
3. Has received radiation therapy or major surgery within 14 days prior to first dose of study drug or has not yet recovered from AEs
4. Has had prior anti-cancer immunotherapy within 4 weeks prior to study intervention, and discontinuation due to grade 3 or 4 toxicities
5. Has ongoing immune-related AEs prior to initiation of study intervention, as defined in the protocol
6. Has known allergy or hypersensitivity to components of the study drug(s)
7. Has any condition requiring ongoing/continuous corticosteroid therapy (>10 mg prednisone/day or anti-inflammatory equivalent) within 1-2 weeks to the first dose of study intervention
8. Has ongoing or recent (within 5 years) evidence of significant autoimmune disease or any other condition that required treatment with systemic immunosuppressive treatments

NOTE: Other Protocol Defined Inclusion / Exclusion Criteria Apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2030-02-03 (Estimated); Study Completion 2030-02-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | Up to Day 29
  Dose escalation
Incidence of Treatment-Emergent Adverse Event (TEAEs) | Approximately 6 Years
  Dose escalation
Incidence of Serious Adverse Events (SAEs) | Approximately 6 Years
  Dose escalation
Incidence of TEAEs leading to treatment discontinuation | Approximately 6 Years
  Dose escalation
Incidence of TEAEs leading to death | Approximately 6 Years
  Dose escalation
Number of participants with Grade 3 laboratory abnormalities | Approximately 6 Years
  Dose escalation Grade 3 or higher per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Objective Response Rate (ORR) per Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria by investigator assessment | Approximately 6 Years
  Dose expansion

SECONDARY OUTCOMES:
ORR based on RECIST 1.1 criteria by investigator assessment | Approximately 6 Years
  Dose escalation
Best Overall Response (BOR) based on RECIST 1.1 criteria | Approximately 6 Years
Duration Of Response (DOR) based on RECIST 1.1 criteria | Approximately 6 Years
Disease control rate based on RECIST 1.1 | Approximately 6 Years
Time to response based on RECIST 1.1 | Approximately 6 Years
Progression Free Survival (PFS) based on RECIST 1.1 | Approximately 6 Years
Concentrations of REGN10597 in serum | Approximately 6 Years
Incidence of Anti-Drug Antibody (ADA) to REGN10597 over time | Approximately 6 Years
Magnitude of ADA to REGN10597 over time | Approximately 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (11):
- United States (11):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Yale School of Medicine, North Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Start Midwest Cancer Research, Grand Rapids, Michigan
  - Northwell Health, Lake Success, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, San Antonio, Texas
  - The Start Center for Cancer Care, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: BrILliance — https://brilliancestudy.com/